CLINICAL TRIAL: NCT03088059
Title: A Pilot Study of Personalized Biomarker-based Treatment Strategy or Immunotherapy in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Biomarker-based Study in R/M SCCHN
Acronym: UPSTREAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1559-HNCG; 2017-000086-74 (EudraCT Number)
Record Dates: First submitted 2017-03-08; First posted 2017-03-23 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Afatinib; palbociclib; Standard of Care; monalizumab; durvalumab; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Patient Cohort B1 (Experimental): Patients who are p16 negative and have an EGFR amplification/mutation or PTEN high or HER2 mutation/amplification will be randomized between afatinib or the standard of care (Methotrexate, Paclitaxel, Docetaxel, Carboplatin, 5-Fluorouracil, Bleomycine, Gemcitabine, Mitomycine or Best supportive care).
  Interventions: Drug: Afatinib; Drug: standard of care
- Patient Cohort B2 (Experimental): Patients who are p16 negative and cetuximab naïve will be randomized between afatinib or the standard of care (Methotrexate, Paclitaxel, Docetaxel, Carboplatin, 5-Fluorouracil, Bleomycine, Gemcitabine, Mitomycine or Best supportive care)
  Interventions: Drug: Afatinib; Drug: standard of care
- Patient Cohort B3 (Experimental): Patients who are p16 negative and have an amplification of CCND1 will be randomized between palbociclib or the standard of care (Methotrexate, Paclitaxel, Docetaxel, Carboplatin, 5-Fluorouracil, Bleomycine, Gemcitabine, Mitomycine or Best supportive care)
  Interventions: Drug: Palbociclib; Drug: standard of care
- Patient Cohort B4 (Experimental): Patients who are p16 negative and 'platinum sensitive' SCCHN will receive niraparib
  Interventions: Drug: Niraparib
- Patient Cohort B5 (Experimental): Patients whith oropharyngeal cancer and which are p16 positive will receive niraparib
  Interventions: Drug: Niraparib
- Patient Cohort I1 (Experimental): Patients who are anti-PD(L)1-naïeve or resistant (primary or secondary resistance) will receive IPH2201 antibody (monalizumab).
  Interventions: Drug: IPH2201
- Patient Cohort I2 (Experimental): Patient who are PD(L)1 pretreated will be randomized between monalizumab + durvalumab or the standard of care (Methotrexate, Paclitaxel, Docetaxel, Carboplatin, 5-Fluorouracil, Bleomycine, Gemcitabine, Mitomycine or Best supportive care)
  Interventions: Drug: standard of care; Drug: IPH2201; Drug: Durvalumab
- Patient Cohort I3 (Experimental): Patient who are progressing prior PD(L)1 after having received at least 2 months of anti-PD(L)-1 will receive INCAGN01876.
  Interventions: Drug: INCAGN01876

INTERVENTIONS:
Drug: Afatinib — Afatinib 40 mg given orally, once daily, 1 cycle is 28 days
  Arms: Patient Cohort B1; Patient Cohort B2
Drug: Palbociclib — Palbociclib 125 mg given orally, once daily, 1 cycle is 28 days (21 days on treatment, then 7 days off)
  Arms: Patient Cohort B3
Drug: standard of care — Methotrexate, Paclitaxel, Docetaxel, Carboplatin, 5-Fluorouracil, Bleomycine, Gemcitabine, Mitomycine or Best supportive care
  Arms: Patient Cohort B1; Patient Cohort B2; Patient Cohort B3; Patient Cohort I2
Drug: IPH2201 — protocol v2.0 and 2.1 : Monalizumab 10mg/kg given intravenously over 60 minutes, once every 14 days, 1 cycle is 14 days protocol v4.0 : Monalizumab 750mg given intravenously over 60 minutes, once every 28 days, 1 cycle is 28 days
  Other Names: Monalizumab
  Arms: Patient Cohort I1; Patient Cohort I2
Drug: Durvalumab — Durvalumab 1500mg given intravenously over 60 minutes, once every 28 days, 1 cycle is 28 days
  Arms: Patient Cohort I2
Drug: Niraparib — Niraparib 300 mg given orally, once daily, 1 cycle is 28 days
  Arms: Patient Cohort B4; Patient Cohort B5
Drug: INCAGN01876 — INCAGN01876 300 mg given intravenously over 30 minutes, once every 14 days, 1 cycle is 28 days
  Arms: Patient Cohort I3

SUMMARY:
This is a biomarker-driven trial that will enroll patients with recurrent or metastatic squamous cell carcinoma of the head and neck progressing after first-line platinum-based chemotherapy. Based on potential biomarkers and molecular alterations identified in the biopsy from the central platform, patients will be allocated in different cohorts. There will be biomarker-positive patient cohorts and immunotherapy cohorts.

ELIGIBILITY:
General Inclusion Criteria:

* Histologically confirmed recurrent and/or metastatic SCCHN of the oral cavity, oropharynx, hypopharynx or larynx not amenable to curative treatment.
* At least one measurable lesion by MRI or CT-scan according to RECIST 1.1, evaluated within 2 weeks prior to registration. Such lesion must not have been previously irradiated; if the measurable lesion(s) have been irradiated, clear progression must be documented.
* Progressive disease after first line platinum-based chemotherapy with or without cetuximab given as palliative treatment or progressive disease within 1 year if platinum-based chemotherapy was given as a part of the multimodal curative treatment. Patients pre-treated with anti-PD1/anti-PDL1 are allowed.
* ECOG performance status 0 -1 with a life expectancy of at least 12 weeks.
* Tumor core biopsy from any accessible tumor at the recurrent or metastatic site available for central testing.
* Patients must have adequate organ function, evaluated within 14 days prior to cohort allocation:
* Hemoglobin ≥ 9 g/100 ml,
* Neutrophils ≥ 1,500/mm3,
* Platelets ≥ 100,000/mm3,
* Total bilirubin <1.5 times the upper limit of normal (ULN) (< 3 times the upper limit of normal for Gilbert's disease),
* Serum ALT and AST ≤ 2.5 x ULN,
* Adequate renal function measured by:
* Estimated creatinine clearance ≥45ml using Cockcroft and Gault formula or Creatinine ≤ 1.5 ULN
* International Normalized Ratio (INR) or Prothrombin Time (PT) must be within the normal ranges as per institution's standard. A window of 5% is allowed.
* Patients receiving anticoagulant therapy are allowed to participate as long as the PT/INR values are within the expected target range of their current dose.
* Clinically normal cardiac function based on -left ventricular ejection fraction (≥ 50%) as assessed either by multi-gated acquisition scan or cardiac ultrasound and 12 lead ECG without clinically relevant abnormalities.
* Patients ≥ 18 years old and must be able to give written informed consent.
* Patients ≥ 70 years old must undergo the G8 screening.
* Women of child-bearing potential must have a negative pregnancy test (serum or urine within the 72 hours prior to cohort allocation).
* Patients of childbearing / reproductive potential must agree to use highly effective methods of contraception based on the Clinical Trial Facilitation Group (CTFG) guidance as of registration and up to 6 months after the last treatment dose. Highly effective methods can achieve failure rate of less than 1% per year when used consistently and correctly. Such methods include: For Women: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal and transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner and sexual abstinence. For Men: condoms, sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient) and no sperm donations during treatment and up to 6 months after last dose of treatment.
* Female subjects who are breast feeding should agree to discontinue nursing prior to the first dose of study treatment and up to 6 months after the last study treatment.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

General Exclusion Criteria:

* Unresolved and significant toxicity CTCAE version 4.03 grade ≥ 2 from previous anticancer therapy other than alopecia.
* History of any of the following cardiovascular conditions within 6 months prior to registration:
* myocardial infarction,
* severe/unstable angina,
* ongoing cardiac dysrhythmias of CTCAE version 4.03 Grade 2 or more,
* atrial fibrillation of any grade,
* coronary/peripheral artery bypass graft,
* symptomatic congestive heart failure according to New York Heart Association (NYHA) Class III or Class IV,
* significant active cardiac disease including uncontrolled high blood pressure defined as systolic ≥150 and diastolic ≥100.
* cerebrovascular accident including transient ischemic attack
* thromboembolic events like symptomatic pulmonary embolism.
* Nasopharynx and sino-nasal tumor.
* Surgery or investigational drugs or chemotherapy or other anticancer therapy within 3 weeks before cohort allocationor or for investigational drugs, within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter. Participant must have recovered from any surgical procedure. Curative radiation therapy (60-70 Gy) within 6 weeks of cohort allocation. Palliative radiation therapy (e.g. 8 Gy on a painful lesion) will be allowed.
* Known untreated and uncontrolled brain metastases or leptomeningeal carcinomatosis.
* Known diagnosis of immune deficiency or a positive serology of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) or pre-existing liver cirrhosis.
* Known pre-existing interstitial lung disease (ILD). Bronchoemphysema is not considered as ILD.
* Other uncontrolled active illnesses or nonmalignant systemic disease (examples include, but are not limited to active infections requiring antibiotics, bleeding disorders, uncontrolled diabetes, uncontrolled ventricular arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome …).
* Any psychiatric, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Any malignancy (other than SCCHN, non-melanoma skin cancer or localized cervical cancer or localized and presumed cured prostatic cancer or basal cell carcinoma of the skin and carcinoma in situ of the cervix or bladder) within the last 3 years prior to treatment allocation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Rate (PFSR) at week 16 | The Progression Free Survival Rate (PFSR) analysis will be performed at week 16 for each patient in cohorts 1, 2 and 3.
  Progression Free Survival Rate (PFSR) at week 16 will be assessed as primary endpoint for all patients from cohorts 1, 2 and 3.
Objective response Rate (ORR) at week 16 | Objective response Rate (ORR) at week 16 will be performed at week 16 for each patient in cohort 4.
  Objective response Rate (ORR) during the first 16 weeks of study treatment will be assessed as primary endpoint for all patients from cohort 4-8.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 54 months after first patient in
Objective Response Rate | 48 months after first patient in
  Objective Response Rate will be measured according to both RECIST 1.1 and iRECIST
Response duration | 54 months after first patient in
Overall Survival (OS) | 54 months after first patient in
Toxicity according CTCAE version 4.03 | 54 months after first patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, for adverse event reporting.
Percentage of patients included in each patient cohort according the biomarker testing | 42 months after first patient in
The percentage of patients with an evaluable fresh tumor biopsy | 42 months after first patient in

CONTACTS AND LOCATIONS:
Locations (33):
- Belgium (11):
  - CHU Saint-Pierre-Site Porte de Hal, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Grand Hopital de Charleroi - Grand Hôpital de Charleroi - Site Notre Dame, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Hopital De Jolimont, Haine-Saint-Paul
  - AZ Groeninge Kortrijk - Campus Kennedylaan, Kortrijk
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - GasthuisZusters Antwerpen - Sint-Augustinus, Wilrijk
  - CHU Dinant Godinne - UCL Namur, Yvoir
- France (9):
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre, Bordeaux
  - Centre Georges-Francois-Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Italy (4):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS - Fondazione G. Pascale, Napoli
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
- Spain (3):
  - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Clinico Universitario De Valencia, Valencia
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust (UHB) - UHB-Queen Elisabeth Medical Centre, Birmingham
  - NHS Lothian - Western General Hospital, Edinburgh
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Guy's and St Thomas' NHS - Guy s and St Thomas' NHS - Guy's Hospital, London
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield

REFERENCES:
- [Derived] Galot R, Le Tourneau C, Guigay J, Licitra L, Tinhofer I, Kong A, Caballero C, Fortpied C, Bogaerts J, Govaerts AS, Staelens D, Raveloarivahy T, Rodegher L, Laes JF, Saada-Bouzid E, Machiels JP. Personalized biomarker-based treatment strategy for patients with squamous cell carcinoma of the head and neck: EORTC position and approach. Ann Oncol. 2018 Dec 1;29(12):2313-2327. doi: 10.1093/annonc/mdy452. PMID 30307465